CLINICAL TRIAL: NCT06376539
Title: Functional Recovery in the First Six Postoperative Months of Cancer Patients Undergoing Lower Limb Resection and Reconstruction. An Observational Study
Brief Title: Functional Recovery of Patients Undergoing Resection and Reconstruction of the Lower Limbs for Bone Tumor.
Acronym: FISIO-ONCO
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CEAVEC: 111/2024/Oss/IOR
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Bone Neoplasm; Rehabilitation
Keywords: bone tumor; physiotherapy; functional recovery
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to describe the course of functional recovery of patients with musculoskeletal tumours and undergone resection and reconstruction operations of lower limbs in the first six months post-surgery, differentiating them on the basis of the anatomical level involved.

DETAILED DESCRIPTION:
Retrospective observational study will be conducted. The evaluation of the patients clinical recovery progress will take place at three different times: during the hospital stay postoperative, at 3 and 6 months after surgery. Different outcome measures will be considered in order to provide a complete picture of the patients functional recovery and their change.

ELIGIBILITY:
Inclusion Criteria:

* All participants undergone lower limb resection and reconstruction with localisation of the disease to the pelvis, femur femur, tibia and foot bones.
* All participants undergone soft tissue resection surgery on the of the lower limb
* All types of oncological diagnoses will be taken considered: osteosarcoma, Ewing and others.

Exclusion Criteria:

* Participants who undergo at our Institute only the surgical treatment while continuing adjuvant treatment at other centres
* Participants for whom no rehabilitation treatment has been activated during adjuvant treatment at our Institute

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants with bone tumor diagnosis treated at the hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Toronto Extremity Salvage Score (TESS) | at 3 months after surgery
  Person's level of independence. It is measured through 30 questions relating to 30 activities of daily living to be answered by the patient. The total score is reported from 0 to 100. A higher score indicates a greater degree of autonomy. A higher score indicates a greater degree of autonomy.
Toronto Extremity Salvage Score (TESS) | at 6 months after surgery
  Person's level of independence. It is measured through 30 questions relating to 30 activities of daily living to be answered by the patient. The total score is reported from 0 to 100. A higher score indicates a greater degree of autonomy. A higher score indicates a greater degree of autonomy.

SECONDARY OUTCOMES:
Range of motion (ROM) | at 3 months after surgery
  The range of motion of the main joints of the lower limbs (hip, knee or foot), measured with a goniometer
Rang of motion - 2 (ROM) | at 6 months after surgery
  The range of motion of the main joints of the lower limbs (hip, knee or foot), measured with a goniometer
Number of participants able to walk | up to 1 week
  Number of participant that are able to walk and aids used for walking
Time Up and Go -2 (TUG) | at 3 months after surgery
  Time it takes a person to get up from a chair, walk three metres, turn around, return to the chair and sit down again is measured.
Time Up and Go (TUG) | at 6 months after surgery
  Time it takes a person to get up from a chair, walk three metres, turn around, return to the chair and sit down again is measured.
Muscle Strength | at 3 months after surgery
  Grades of Muscle Strength from 0 (no contraction) to 5 (best strength)
Muscle Strength-2 | at 6 months after surgery
  Grades of Muscle Strength from 0 (no contraction) to 5 (best strength)
Number of day from surgery to first walking | up to 1 week
  The number of day that participants needs to recover ambulation after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morri M, Venturini E, Abbruzzese A, Meneghini M, Raffa D, Berti L, Donati D. The functional recovery trajectory in patients undergoing lower limb salvage surgery for bone tumour: an observational study. Support Care Cancer. 2026 Jan 28;34(2):136. doi: 10.1007/s00520-026-10374-x. PMID 41593389